CLINICAL TRIAL: NCT02700100
Title: Prospective, Non-randomised, Open Label Clinical Study to Assess the Safety of the Bioabsorbable Pulmonary Valved Conduit (PV-001) in Subjects Undergoing Right Ventricular Outflow Tract (RVOT) Reconstruction
Brief Title: Study to Assess Safety of the Pulmonary Valved Conduit (PV-001) in Subjects Undergoing Right Ventricular Outflow Tract Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-01
Record Dates: First submitted 2016-02-15; First posted 2016-03-07 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulmonary Valved Conduit (PV-001) (Experimental): Bioabsorbable Pulmonary Valved Conduit (PV-001) implantation through open surgery.
  Interventions: Device: Bioabsorbable Pulmonary Valved Conduit (PV-001)

INTERVENTIONS:
Device: Bioabsorbable Pulmonary Valved Conduit (PV-001) — The Bioabsorbable Pulmonary Valved (PV) Conduit (PV-001) is a polymer-based medical device, with a total length of 8 cm with inner diameters of 16 or 18 mm. The valve itself is formed by three leaflets, incorporated within the conduit wall.
  The PV conduit is used for correction or reconstruction of the Right Ventricular Outflow Tract (RVOT) in patients with any of the following congenital heart malformations:
  * Tetralogy of Fallot
  * Truncus Arteriosus
  * Pulmonary Atresia
  * Transposition of Great Arteries with Ventricular Septal Defect (VSD)
  * Pulmonary Stenosis in combination with other defects in congenital heart defect (CHD) syndromes
  The PV conduit can also be used for replacement of previously implanted, but dysfunctional, pulmonary homografts or valved conduits.

SUMMARY:
The study is a prospective, non-randomised, open label clinical study to assess the safety of the Bioabsorbable Pulmonary Valved (PV) conduit (PV-001) in subjects > 2 years and < 22 years of age, undergoing Right Ventricular Outflow Tract (RVOT) reconstruction. It is a first in man feasibility study which will include 10-12 patients in up to 6 sites in Europe.

The primary objective of the study is to assess the survival rate of subjects at 6 months following implantation of the Bioabsorbable Pulmonary Valved Conduit (PV-001).

Secondary objectives:

1. The survival rate of subjects at 12 months following implantation of the Bioabsorbable Pulmonary Valved Conduit (PV-001)
2. The percentage of conduit failure at 6 months and 12 months, where conduit failure includes the need for reintervention or reoperation.
3. The pressure gradient across the pulmonary valve will have an acceptable level at 12 months follow up.
4. The pulmonary regurgitation measured will not exceed a moderate grading at 12 months follow up.
5. To evaluate the usability of the Bioabsorbable Pulmonary Valved Conduit (PV-001) during the surgical procedure, using exploratory parameters

Long term safety will be assessed up to 60 months post implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring RVOT reconstruction, suitable for 16 mm or 18 mm conduit.
2. Male or Female.
3. Age > 2 years and < 22 years.
4. Right Ventricular to Pulmonary Artery peak gradient > 35mm Hg or moderate or severe Pulmonary Valve regurgitation (≥3+), or have both.
5. The patient, and the patient's parent / legal representative where appropriate, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent by signing the approved informed consent form.
6. The patient, and the patient's parent / legal representative where appropriate, and the treating physician agree that the subject will return for all required post-procedure follow up visits and the subject will comply with protocol-required follow-up visits.

Exclusion Criteria:

1. Need for or presence of prosthetic valve at other position.
2. Need for concomitant surgical procedures (outside of the heart).
3. Patients with previously implanted pacemaker (including defibrillators), or mechanical valves.
4. Active infection requiring current antibiotic therapy (if temporary illness, subject may be a candidate 4 weeks after discontinuation of antibiotics).
5. Active endocarditis.
6. Leukopenia.
7. Acute or chronic anaemia.
8. Thromocytopenia.
9. Severe chest wall deformity.
10. Right ventricular outflow tract aneurysm.
11. Known hypersensitivity to anticoagulants and antiplatelet drugs.
12. Immunocompromised patient defined as: autoimmune disease, patients receiving immunosuppressant drugs or immunostimulant drugs.
13. Need for emergency cardiac or vascular surgery or intervention.
14. Major or progressive non-cardiac disease (liver failure, renal failure, cancer) that has a life expectancy of less than one year.
15. Currently participating, or participated within the last 30 days, in an investigational drug or device study.
16. Alcohol or drug abuse as defined by DSM IV-TR criteria for substance abuse - this includes the illicit use of cannabis within the last 12 months.
17. Pregnancy.
18. Females who are sexually active and are not willing to use adequate contraceptive precautions for the next 2 years
19. Subject has medical, social or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
The survival rate of participants at 6 months following implantation of the Bioabsorbable Pulmonary Valved Conduit (PV-001),, measured by the fact that the patient is still alive at the time of the 6 month FU visit | 6 months

SECONDARY OUTCOMES:
The survival rate of participants at 12 months following implantation of the Bioabsorbable Pulmonary Valved Conduit (PV-001), measured by the fact that the patient is still alive at the time of the 12 month FU visit. | 12 months
The rate of reoperation or reintervention due to PV conduit failure at 6 months and 12 months follow up , measured by the fact that the patient did not have a reoperation or reintervention during the follow up time. | 6 and 12 months
The rate of patients with a mean pressure gradient across the area of PV conduit implantation (RV to PA) of less than 40 mm Hg at 12 months follow up, measured with echocardiography at 12 months follow up. | 12 months
The rate of patients with pulmonary regurgitation of equal or less than moderate at 12 months follow up, measured with echocardiography at 12 months follow up. | 12 months
  The degree of pulmonary regurgitation (the percentage of blood that regurgitates back through the pulmonary valve due to valve insufficiency) is defined as:
  * mild if regurgitant fraction is <20%
  * moderate if regurgitant fraction is 20%-40%;
  * severe if regurgitant fraction is >40%.
Overall satisfaction of the implantability of the Bioabsorbable Pulmonary Valved Conduit (PV-001), measured with a questionnaire given to the implanting surgeon at the time of implantation of the PV conduit (PV-001). | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Carrel, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (3):
- Gottsegen György Hungarian Institute of Cardiology, Paediatric Cardiac Centre, Budapest, Hungary
- Institute Jantung Negara, National Heart Institute, Kuala Lumpur, Malaysia
- University Children's Hospital of Cracow (UCH),, Krakow, Poland

REFERENCES:
- [Derived] Morales DL, Herrington C, Bacha EA, Morell VO, Prodan Z, Mroczek T, Sivalingam S, Cox M, Bennink G, Asch FM. A Novel Restorative Pulmonary Valve Conduit: Early Outcomes of Two Clinical Trials. Front Cardiovasc Med. 2021 Mar 4;7:583360. doi: 10.3389/fcvm.2020.583360. eCollection 2020. PMID 33748192